CLINICAL TRIAL: NCT03073330
Title: One vs Two Step Approach for GDM Screening
Brief Title: One Step Versus Two Step Approach for Gestational Diabetes Mellitus Screening
Acronym: OTSAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, adeeb khalifeh, Physician Fellow, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8550
Record Dates: First submitted 2016-08-11; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One Step (Experimental): The intervention is gestational diabetes screening with 2 hour GTT 75 g load.
  Interventions: Diagnostic Test: GDM screening with 75 g 2 hour GTT
- Two Step (Active Comparator): There is no intervention is this arm as patients will subjected to routine gestational diabetes screening with one hour glucola, 50 g load.
  Interventions: Diagnostic Test: GDM screening with two step approach

INTERVENTIONS:
Diagnostic Test: GDM screening with 75 g 2 hour GTT — Patients will be diagnosed with gestational diabetes if they have one abnormal value: Fasting ≥ 92; 2 hour ≥ 180 mg/dl;1 hour ≥ 153 mg/dl.
  Arms: One Step
Diagnostic Test: GDM screening with two step approach — 1 hour glucola with 50 g glucose load followed by 100 g glucose load if 1 hour glucola positive
  Arms: Two Step

SUMMARY:
Our study will assess if there is a difference in incidence of gestational diabetes using different screening approaches, either using a one-step approach with a 2 hour glucose tolerance test or using a two-step approach. Prior studies have proven similar incidences including a randomized controlled trial.

DETAILED DESCRIPTION:
Gestational Diabetes is screened for in pregnancy by drinking a solution containing a certain amount of glucose and testing blood glucose level one hour after drinking it. If this value is above a certain cut-off (>135mg/dl), the patient is subjected to another test involving drinking a solution containing a higher amount of glucose and checking blood glucose while fasting, 1 hour after drinking the solution and 2 hours after drinking the solution. (Two step approach).

Cut off values will be: 3 hour>180 mg/dl, 2 hour > 155 mg/dl, 1hour >140 mg/dl, fasting >95mg/dl. Two abnormal values will meet the diagnosis of gestational diabetes.

In other parts of the United States, and most of the rest of the word, screening for gestational diabetes uses a one-step approach by drinking a solution containing 75g of glucose (As recommended by the American Diabetic Society, the Endocrine Society, WHO and the International Association of Diabetes and Pregnancy Study groups1-3). Blood glucose values are checked at fasting, one hour and two hours after solution drinking.

The diagnosis of gestational diabetes is based on one elevated values. (cut off: Fasting ≥92mg/dl, 1hour ≥180 mg/dl, 2 hours ≥153 mg/dl).

Our study will assess if there is a difference in incidence of gestational diabetes using these different screening approaches. Prior studies have proven similar incidences including a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 16-50 year of age
* Pregnant women (limits the participants to female gender)

Exclusion Criteria:

* Pregestational Diabetes Mellitus
* History of bariatric surgery

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women (limits the participants to female gender)
Enrollment: 284 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of gestational diabetes diagnosed on each screening test of each arm. | at the time of the screening
  Gestational diabetes will be made based on one abnormal value. Fasting ≥126 mg/dl; 1 hour≥ 180 mg/dl and 2 hour ≥ 153 mg/dl

SECONDARY OUTCOMES:
neonatal hyperbilirubinemia | first 48 hours of life
  incidence of neonatal hyperbilirubinemia
mode of delivery | at time of delivery
  incidence of cesarean delivery, spontaneous vaginal delivery, operative vaginal delivery, and induction of labor
gestational age at delivery | at time of delivery
  gestational age at delivery
Anal sphincter injury | at time of delivery
  Incidence of Anal sphincter injury
Shoulder dystocia | at time of delivery
  incidence of shoulder dystocia, and birth trauma
Neonatal complications | between birth and 28 days of age
  includes necrotizing enterocolitis, respiratory distress syndrome, intraventricular hemorrhage, hypoglycemia, jaundice, hyperbilirubinemia, perinatal death, admission to neonatal intensive care unit
Hypertensive disorders in pregnancy | 6 months
  includes gestational hypertension, preeclampsia
Fetal growth restriction, large for gestational age and polyhydramnios | 6 months
  Incidence of Fetal growth restriction,large for gestational age and polyhydramnios
Birth weight | Time of delivery
  Mean of birth weight and incidence of macrosomia
Apgar score | at 1, 5 and 10 minutes after birth
  Apgar score

CONTACTS AND LOCATIONS:
Overall Officials: Adeeb Khalifeh, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Southwick AM, Wang LX, Long SR, Lee YC. Activity of Sinorhizobium meliloti NodAB and NodH enzymes on thiochitooligosaccharides. J Bacteriol. 2002 Jul;184(14):4039-43. doi: 10.1128/JB.184.14.4039-4043.2002. PMID 12081977